CLINICAL TRIAL: NCT03560492
Title: A Comparative Study of Postural Garment Versus Exercises for Women With Non-specific Cervical Pain: a Randomised Crossover Trial.
Brief Title: Postural Garment Versus Exercises for Women With Cervical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Andorra (Other)
Responsible Party: Principal Investigator, Merce AVELLANET, Head of Rehabilitation Department - Adjunct professor, University of Andorra
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UA001GRCSSS
Record Dates: First submitted 2018-05-03; First posted 2018-06-18 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Posture; Cervical Pain
Keywords: posture; cervical pain; exercise
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomised to receive one intervention during the initial 3 month phase of the study and receive the other intervention during the second 3 month phase of the study, after a wash out 3 month period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Postural assessment is performed by a blinded investigator with a device for computerized measurement of surface curvature in the upright position (SpinalMouse®).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posture Plus Force (Experimental): Participants are provided with the posture garment. They have to wear it 2 to 4 h per day for a 3 month period. Participants receive a logbook that should be filled every day.
  Interventions: Device: Posture garment
- Exercise (Active Comparator): A physiotherapist teaches exercises to participants (5 sessions of 20 minutes each of stretching and strengthening exercises). Exercises are focused on cervical and dorsal areas, Participants receive instructions to continue at home on a daily basis for 3 months. Participants receive a logbook that should be filled every day.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — 5 sessions of exercises of 20 minutes each. Participants have to do a set of cervical, dorsal and abdominal stretching and strengthening exercises. Participants receive instructions to continue at home on a daily basis for 3 months and record compliance in a logbook.
  Arms: Exercise
Device: Posture garment — Participants are provided with the appropriate size of a posture garment which includes thoracic and abdominal tensional bands. They are instructed to wear it 2 to 4 h per day for a 3 month period and record compliance in a logbook daily.
  Arms: Posture Plus Force

SUMMARY:
This study aim to compare a new postural garment (Posture Plus Force ®) versus exercises in women with non specific cervical pain. The investigators focus on nurses and allied health professionals due to the importance of posture in work related musculoskeletal disorders.

DETAILED DESCRIPTION:
OBJECTIVE: To investigate the effects of a postural garment versus exercises in nurses with non-specific cervical pain.

DESIGN: Randomized cross over clinical trial with a 3 months sequence treatment and a 3 months washout period..

PARTICIPANTS: Nurses and allied health professionals with cervical pain aged 21 to 55 years.

INTERVENTIONS:

Participants are allocated at random to receive interventions in two groups:

* P+ : a postural garment (Posture Plus Force - FGP srl ® - Italy) to be worn from 2 to 4 hours per day, during 90 days.
* Ex: five physiotherapy sessions to learn stretching and strengthening exercises (20 minutes) with instructions to continue at home on a daily basis for 90 days.

The subjects in each group will be cross over after three months of wash out period.

MAIN OUTCOME MEASURES:

The primary outcomes are postural control and pain intensity. Pictures on sagittal and frontal plane as well as measurements of static posturography with a scan (SpinalMouse ®) are conducted at T0 (pre-intervention), T1 immediately after garment fitting for P+ group and after the 5th session for Ex group, T30, T60 and T90 at day 30, day 60 and day 90 of follow-up. Pain is measured by visual analogue scale (VAS) on the same assessment days.

STATISTICAL ANALYSIS:

Statistical analysis is conducted following intention-to-treat principles, and the treatment effects calculated using linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Nurses and health allied professionals females with cervical pain
* Voluntarily signed informed consent
* Able to wear the garment and to do exercises and follow up assessments

Exclusion Criteria:

* Pregnancy
* Malignancy or other severe disease
* Cervical pain with significant extremity symptoms and/or neurological dysfunction (cervical radiculopathy and cervical spondylotic myelopathy)
* Unable to perform exercises
* Unwilling to do follow up assessments
* Psychiatric disorders

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline cervical Pain measured with a visual analog scale at 3 months | Pain is assessed pre-intervention (Day 0) and at Month 3 of follow-up.
  Visual analogue scale is a psychometric measuring instrument designed to document cervical pain severity in individual subjects. It achieves a rapid (statistically measurable and reproducible) classification of symptom severity. A 100-mm long horizontal line with verbal descriptors is used to grade the amount of pain that a patient feels from no pain (left 0 mm) to an extreme amount of pain (right 100 mm).
Change from baseline cervical Pain at 3 months (after the wash out period) | After the washout period, pain is assessed at baseline (Month 6) and after 3 months of intervention (Month 9)
  Visual analogue scale is a psychometric measuring instrument designed to document cervical pain severity in individual subjects. It achieves a rapid (statistically measurable and reproducible) classification of symptom severity. A 100-mm long horizontal line with verbal descriptors is used to grade the amount of pain that a patient feels from no pain (left 0 mm) to an extreme amount of pain (right 100 mm).

SECONDARY OUTCOMES:
Posture measured by angle of Kyphosis and angle of lordosis with a computerized device (SpinalMouse® ) | Posture is assessed pre-intervention (Day 0))
  SpinalMouse ® is a device that, combined with a computer program, assesses the curvatures of the spine without applying radiation. The device is guided manually on the skin along the spinous process apophysis from C7 to S3. The measuring head follows their contour in the sagittal plane and records clinically relevant data. A software program using an algorithm uses this information to calculate the angle of kyphosis and angle of lordosis. Data obtained have been proved to be reliable and accurate
Posture measured by angle of Kyphosis and angle of lordosis with a computerized device (SpinalMouse® ) | Posture is assessed at Month 3 of follow-up.
  SpinalMouse ® is a device that, combined with a computer program, assesses the curvatures of the spine without applying radiation. The device is guided manually on the skin along the spinous process apophysis from C7 to S3. The measuring head follows their contour in the sagittal plane and records clinically relevant data. A software program using an algorithm uses this information to calculate the angle of kyphosis and angle of lordosis. Data obtained have been proved to be reliable and accurate
Posture measured by angle of Kyphosis and angle of lordosis with a computerized device (SpinalMouse® ) | Posture measurement is repeated after the 3-month washout period (Month 6)
  SpinalMouse ® is a device that, combined with a computer program, assesses the curvatures of the spine without applying radiation. The device is guided manually on the skin along the spinous process apophysis from C7 to S3. The measuring head follows their contour in the sagittal plane and records clinically relevant data. A software program using an algorithm uses this information to calculate the angle of kyphosis and angle of lordosis. Data obtained have been proved to be reliable and accurate
Posture measured by angle of Kyphosis and angle of lordosis with a computerized device (SpinalMouse® ) | Posture is assessed at Month 9 (end of study) after the washout period and the cross over 3 months intervention
  SpinalMouse ® is a device that, combined with a computer program, assesses the curvatures of the spine without applying radiation. The device is guided manually on the skin along the spinous process apophysis from C7 to S3. The measuring head follows their contour in the sagittal plane and records clinically relevant data. A software program using an algorithm uses this information to calculate the angle of kyphosis and angle of lordosis. Data obtained have been proved to be reliable and accurate
Neck Disability Index | Neck disability is assessed pre-intervention (Day 0)
  Cervical pain-related disability will be assessed with the validated Spanish version of Neck Disability Index. The Neck Disability Index is a ten-item questionnaire based on the Oswestry Low Back Pain Index that assesses disability associated with neck pain and whiplash. There are four items that relate to subjective symptomatology (pain intensity, headache, concentration, sleeping) and six items that relate to activities of daily living (lifting, work, driving, recreation, personal care, reading). The questionnaire is self and administered requires only 5-10 minutes to complete. It is scored from 0 (no disability) to 50 (maximum disability). Each subject select from one of six potential responses for each item ranging from no disability (0) to total disability (5). The ten items are summed to gain the total score.
Neck Disability Index | Neck disability is assessed at Month 3 of follow-up.
  Cervical pain-related disability will be assessed with the validated Spanish version of Neck Disability Index. The Neck Disability Index is a ten-item questionnaire based on the Oswestry Low Back Pain Index that assesses disability associated with neck pain and whiplash. There are four items that relate to subjective symptomatology (pain intensity, headache, concentration, sleeping) and six items that relate to activities of daily living (lifting, work, driving, recreation, personal care, reading). The questionnaire is self and administered requires only 5-10 minutes to complete. It is scored from 0 (no disability) to 50 (maximum disability). Each subject select from one of six potential responses for each item ranging from no disability (0) to total disability (5). The ten items are summed to gain the total score.
Neck Disability Index | Neck disability is repeated after the 3-month washout period (Month 6)
  Cervical pain-related disability will be assessed with the validated Spanish version of Neck Disability Index. The Neck Disability Index is a ten-item questionnaire based on the Oswestry Low Back Pain Index that assesses disability associated with neck pain and whiplash. There are four items that relate to subjective symptomatology (pain intensity, headache, concentration, sleeping) and six items that relate to activities of daily living (lifting, work, driving, recreation, personal care, reading). The questionnaire is self and administered requires only 5-10 minutes to complete. It is scored from 0 (no disability) to 50 (maximum disability). Each subject select from one of six potential responses for each item ranging from no disability (0) to total disability (5). The ten items are summed to gain the total score.
Neck Disability Index | Neck disability is assessed at Month 9 (end of study) after the washout period and the cross over 3 months intervention
  Cervical pain-related disability will be assessed with the validated Spanish version of Neck Disability Index. The Neck Disability Index is a ten-item questionnaire based on the Oswestry Low Back Pain Index that assesses disability associated with neck pain and whiplash. There are four items that relate to subjective symptomatology (pain intensity, headache, concentration, sleeping) and six items that relate to activities of daily living (lifting, work, driving, recreation, personal care, reading). The questionnaire is self and administered requires only 5-10 minutes to complete. It is scored from 0 (no disability) to 50 (maximum disability). Each subject select from one of six potential responses for each item ranging from no disability (0) to total disability (5). The ten items are summed to gain the total score.
Pain Catastrophizing Scale | Assessed pre-intervention (Day 0)
  In order to assess the catastrophizing dimension related to pain, the Pain Catastrophizing Scale is used. It is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time) that yields a total score and three subscale scores assessing rumination, magnification and helplessness. Total score ranges from 0 to 52. It is a self-report measurement tool that provided a valid index of catastrophizing in clinical populations.
Pain Catastrophizing Scale | Assessed at Month 3 of follow-up.
  In order to assess the catastrophizing dimension related to pain, the Pain Catastrophizing Scale is used. It is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time) that yields a total score and three subscale scores assessing rumination, magnification and helplessness. Total score ranges from 0 to 52. It is a self-report measurement tool that provided a valid index of catastrophizing in clinical populations.
Pain Catastrophizing Scale | Pain Catastrophizing scale is repeated after the 3-month washout period (Month 6)
  In order to assess the catastrophizing dimension related to pain, the Pain Catastrophizing Scale is used. It is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time) that yields a total score and three subscale scores assessing rumination, magnification and helplessness. Total score ranges from 0 to 52. It is a self-report measurement tool that provided a valid index of catastrophizing in clinical populations.
Pain Catastrophizing Scale | Catastrophizing is assessed at Month 9 (end of study) after the washout period and the cross over 3 months intervention
  In order to assess the catastrophizing dimension related to pain, the Pain Catastrophizing Scale is used. It is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time) that yields a total score and three subscale scores assessing rumination, magnification and helplessness. Total score ranges from 0 to 52. It is a self-report measurement tool that provided a valid index of catastrophizing in clinical populations.

OTHER OUTCOMES:
Garment comfort | garment comfort is assessed at Month 1 when allocated to the garment group intervention.
  Garment comfort is evaluated with a 5-point Likert scale with the following anchors • 1 - Very dissatisfied • 2 - dissatisfied • 3 - unsure • 4 - satisfied • 5 - Very satisfied
Garment comfort | garment comfort is assessed at Month 3 when allocated to the garment group intervention.
  Garment comfort is evaluated with a 5-point Likert scale with the following anchors • 1 - Very dissatisfied • 2 - dissatisfied • 3 - unsure • 4 - satisfied • 5 - Very satisfied
Assessment of global perceived effect of treatment | Perceived effect of treatment is assessed at Month 3 of follow-up.
  Assessment of global perceived effect of treatment is performed with a Visual Analog Scale . Visual analogue scale is a psychometric measuring instrument designed to document perceived effect of the treatment in individual subjects. A 100-mm long horizontal line with verbal descriptors is used to grade the perceived effect that a patient feels from no improvement (left 0 mm) to an great improvement (right 100 mm).
Assessment of global perceived effect of treatment | Perceived effect of treatment is assessed at Month 9 (end of study)
  Assessment of global perceived effect of treatment is performed with a Visual Analog Scale . Visual analogue scale is a psychometric measuring instrument designed to document perceived effect of the treatment in individual subjects. A 100-mm long horizontal line with verbal descriptors is used to grade the perceived effect that a patient feels from no improvement (left 0 mm) to an great improvement (right 100 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Merce Avellanet, MD, PhD, Principal Investigator — Universitat d'Andorra
Locations (1):
- Hospital N Sra de Meritxell - Rehabilitation Department, Les Escaldes, Spanish, Andorra

REFERENCES:
- [Derived] Avellanet M, Boada-Pladellorens A, Perrot JC, Loro L, Rodrigo Cansado L, Monterde D, Romagosa J, Gea E. Comparative Study of Postural Garment Versus Exercises for Patients With Nonspecific Cervical Pain: Protocol for a Randomized Crossover Trial. JMIR Res Protoc. 2020 Apr 16;9(4):e14807. doi: 10.2196/14807. PMID 32297876